CLINICAL TRIAL: NCT04663373
Title: Prognostic Impact of Physical Activity Patterns After Percutaneous Coronary Intervention - The PIPAP Observational Study
Brief Title: Prognostic Impact of Physical Activity Patterns After Percutaneous Coronary Intervention (PIPAP Study)
Acronym: PIPAP
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: ID 2020-01861
Record Dates: First submitted 2020-11-19; First posted 2020-12-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Physical Activity; Coronary Artery Disease
Keywords: Step counting; Accelerometer; Percutaneous coronary intervention; Risk prediction; Major adverse cardiac event
MeSH Terms: conditions — Motor Activity; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Step counting — Patients are given a physical activity tracker (wrist band) that they are asked to wear for two weeks after discharge from percutaneous coronary intervention.

SUMMARY:
Physical activity monitoring after coronary bypass grafting and other major surgeries has been found to be predictive for hospital readmission and adverse outcome. In patients after percutaneous coronary intervention (PCI) it has been found that a patient reported activity score is predictive of 3 year major adverse coronary event (MACE). It is not known whether physical activity shortly after discharge from PCI is predictive of one-year MACE. Early identification of patients at increased risk of MACE would facilitate the intensification of preventive strategies in these patients.

Primary objective is the quantification of physical activity (daily steps) during the first two weeks after hospital discharge as a predictor for MACE at one year. Secondary objectives are: 1) Comparison between daily steps and objectively measured activity counts (divided in time spent in moderate-to-vigorous activity, light activity and sedentary activity), as well as patient reported activity; 2) Association of daily steps after one year with reaching targets for systolic blood pressure, low-density lipoprotein cholesterol (LDL-C), body mass index (BMI) and glycated haemoglobin (HbA1c); 3) Comparison of daily steps after hospital discharge and MACE between non cardiac rehabilitation (CR), conventional hospital based CR, tele-CR and modular CR participants; 4) Comparison of daily steps at one year after hospital discharge in different CR groups.

DETAILED DESCRIPTION:
Study design

This is a monocentric open label explorative study (with primary objective to assess the predictive value of daily steps for MACE). Patients will be asked to wear an activity tracker for two weeks following hospital discharge. Patients who participate in any form of CR in our institution and attend the routine check-up 12 month after PCI in our institution will be asked to wear the activity tracker again for two weeks.

Study intervention

Patients will be informed about the study by the prevention team (advanced nurse practitioners) usually on the day of discharge from PCI during the routine visit by this team to inform patients about the different options of CR. Patients will be provided with an activity tracker in the form of a wrist band, the patient information sheet including informed consent (IC), the International Physical Activity Questionnaires Short-Form (IPAQ-SF) and an addressed and prepaid envelope. They are asked to read the patient information when arrived at home, sign the IC when willing to participate and wear the wrist band continuously for two weeks after hospital discharge. After that, they should send the wrist band, the filled in IPAQ-SF and signed IC in the provided envelope to our institute. If they are unwilling to participate, they can send the activity tracker back straight away. Patients attending the clinical routine check-up after 12 months in our institution will be asked to wear the activity tracker again for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for ambulatory cardiac rehabilitation (CR, patients not living in nursing home, not enrolling in stationary CR)
* Signing informed consent

Exclusion Criteria:

* Staged PCI;
* Previous participation in this study;
* Inability or contraindications to undergo CR (nursing home residence, stationary CR, orthopedic or neurologic impairment prohibiting physical exercise, psychiatric conditions)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc..

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated by percutaneous coronary intervention at the University Clinic of Cardiology, University Hospital Bern, Berne, Switzerland. Consecutive patients who are eligible for ambulatory CR are seen by the prevention team (nurse practitioners) usually on the day of hospital discharge from PCI and will be informed about the different forms of CR and the study.
Sampling Method: Non-Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event | One year
  Major Adverse Cardiac Events (MACE) at one year after percutaneous coronary intervention

SECONDARY OUTCOMES:
Number of steps | One year
  Number of steps per day will be measured during the first two weeks after Hospital discharge. Mean steps per day over the two weeks wearing time will be related to MACE at one year.
Time spent with moderate to high intensity activity per day | One year
  Physical activity will be measured during the first two weeks after Hospital discharge and association with MACE at one year will be tested
Sedentary time | One year
  Sedentary time will be measured during the first two weeks after Hospital discharge and association with MACE at one year will be tested
Changes in number of daily steps | One year
  Changes in number of steps during the two weeks of tracker wearing time will be measured during the first two weeks after Hospital discharge and association with MACE at one year will be tested
Changes in volume of daily physical activity | One year
  Predictors for changes in volume of daily physical activity during the two weeks after Hospital discharge will be sought from anthropometric Parameters, medical history, cardiovascular Risk factors, socioeconomic Parameters, completion of cardiac rehabilitation by multivariate regression analysis
Identification of predictors of number of steps | One month
  Predictors of steps during the two weeks after Hospital discharge will be sought from anthropometric Parameters, medical history, cardiovascular Risk factors, socioeconomic Parameters, completion of cardiac rehabilitation by multivariate regression analysis
Identification of predictors of physical activity | One month
  Predictors of physical activity during the two weeks after Hospital discharge will be sought from anthropometric Parameters, medical history, cardiovascular Risk factors, socioeconomic Parameters, completion of cardiac rehabilitation by multivariate regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Wilhelm, MD, Study Chair — Preventive Cardiology & Sports Medicine; Eser Prisca, PhD, Study Director — Preventive Cardiology & Sports Medicine
Locations (1):
- Department of Preventive Cardiology, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data sharing plan is not yet Ready, patient daily step Counts will be made available to other Researchers together with main clinical patient data.
Time Frame: not yet decided
Access Criteria: not yet decided

REFERENCES:
- [Derived] Gonzalez-Jaramillo N, Eser P, Casanova F, Bano A, Franco OH, Windecker S, Raber L, Wilhelm M. Prognostic impact of physical activity patterns after percutaneous coronary intervention. Protocol for a prospective longitudinal cohort. The PIPAP study. Front Cardiovasc Med. 2022 Sep 30;9:976539. doi: 10.3389/fcvm.2022.976539. eCollection 2022. PMID 36247455
- [Derived] Eser P, Gonzalez-Jaramillo N, Weber S, Fritsche J, Femiano R, Werner C, Casanova F, Bano A, Franco OH, Wilhelm M. Objectively measured adherence to physical activity among patients with coronary artery disease: Comparison of the 2010 and 2020 World Health Organization guidelines and daily steps. Front Cardiovasc Med. 2022 Sep 28;9:951042. doi: 10.3389/fcvm.2022.951042. eCollection 2022. PMID 36247452

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT04663373/SAP_000.pdf